CLINICAL TRIAL: NCT00124358
Title: An Evaluation of Innovative Methods for Integrating Buprenorphine Opioid Treatment in HIV Primary Care Settings
Brief Title: Buprenorphine and Integrated HIV Care Evaluation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The New York Academy of Medicine (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency); El Rio Santa Cruz Neighborhood Health Center (Unknown); Organization to Achieve Solutions in Substance Abuse (OASIS) (Other); Oregon Health and Science University (Other); Montefiore Medical Center (Other); University of Miami (Other); Brown University (Other); University of California, San Francisco (Other); Johns Hopkins University (Other); CORE Center, Cook County Bureau of Health Services (Unknown); Yale University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 063005; H97HA03795
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2007-03-27 (Estimated); Status verified 2007-03

CONDITIONS: Opioid-Related Disorders; HIV Infections; AIDS
Keywords: Drug Abuse; Drug Addiction; Drug Dependence; Drug Use Disorders; Drug Use Disorder; Substance Abuse; Substance Use Disorder; Buprenorphine; Opiate Addiction; Substance-related disorders; HIV
MeSH Terms: conditions — Opioid-Related Disorders; HIV Infections; Acquired Immunodeficiency Syndrome; Substance-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine
Behavioral: Integrated HIV care and office-based opioid dependence treatment

SUMMARY:
The purpose of this study is to assess the feasibility, cost and effectiveness of interventions designed to integrate buprenorphine treatment for opioid dependence into HIV primary care in ten HIV care centers in the U.S.

DETAILED DESCRIPTION:
Programs that integrate medical care and drug treatment have shown great promise in improving health and substance use related outcomes. The overlap in the epidemics of HIV (with its complex medical needs) and drug abuse makes HIV-infected drug users a population likely to benefit from the integration of primary care and drug treatment. The Drug Addiction Treatment Act of 2000 and the approval of buprenorphine for the office-based treatment of opioid addiction provide a new opportunity to integrate addiction treatment and medical care for people with HIV. Research has demonstrated the effectiveness of buprenorphine in reducing illicit drug use among opioid dependent people. However, little is known about implementing such programs in HIV care settings, their cost, what effect they have on the health outcomes and substance use behavior of PLWH/A, or their broader impact on providers, institutions, and local systems.

Through this study, approximately 1,350 HIV-infected individuals who meet criteria for opioid dependence will be selected by eleven model demonstration projects located in ten HIV care centers across the U.S. Information on patients' drug use, HIV health status, service utilization, quality of life, and satisfaction with services as well as information about providers' practices and attitudes towards treating drug dependent patients will be collected through face-to-face interviews, audio computer-assisted self-interviewing, written surveys, and chart abstractions. These data will be used to help replicate effective programs that integrated HIV care and drug treatment and to improve the care of HIV-infected opioid dependent individuals.

Comparisons: All eleven programs will compare a group of patients who receive integrated buprenorphine treatment and HIV care to a group of patients who receive an alternate intervention. However, the program designs and comparison group interventions vary across the sites and are locally determined. Some sites will implement randomized control designs, while others will use observational methods.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Clinical diagnosis of opioid dependence
* Fluent in English or Spanish
* 18 years or older

Exclusion Criteria:

* Liver function tests (transaminase only) at five times or higher than normal level;
* Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition (DSM-IV) criteria for benzodiazepine abuse or dependence within the past 6 months;
* DSM-IV criteria for alcohol dependence within the past 6 months;
* Actively suicidal;
* Psychiatric impairment that impedes ability to consent (dementia, delusional, actively psychotic);
* Methadone dose exceeding levels allowing for safe transition to buprenorphine;
* Pregnant women and women actively trying to become pregnant;
* Clinical judgment of local site principal investigator that patient is inappropriate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1350
Dates: Start 2005-08; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Substance use outcomes at 1, 3 and 6 months measured by self-report
Urine toxicology results at 1, 3, 6, and 12 months
Retention in and adherence to HIV care at 1, 3, 6, and 12 months

SECONDARY OUTCOMES:
Quality of life at 1, 3, 6, 9, and 12 months
HIV-related health outcomes at 1, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Finkelstein, ScD, Principal Investigator — New York Academy of Medicine; David Fiellin, MD, Principal Investigator — Yale University
Locations (10):
- United States (10):
  - El Rio Santa Cruz Neighborhood Health Center, Tucson, Arizona
  - Organization to Achieve Solutions in Substance Abuse, Oakland, California
  - University of California San Francisco, San Francisco, California
  - Yale University School of Medicine AIDS Program, New Haven, Connecticut
  - University of Miami School of Medicine, Miami, Florida
  - The CORE Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Montefiore Medical Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - The Miriam Hospital, Providence, Rhode Island

REFERENCES:
- See also: Click here for more information about this study: Buprenorphine and Integrated HIV Care Evaluation and Support Center (BHIVES). — http://www.bhives.org